CLINICAL TRIAL: NCT01028924
Title: A Randomised, 4-period, Placebo and Active-controlled, Single-dose, Change-over Trial to Evaluate the Effects of Teduglutide on Cardiac Repolarisation and Conduction in Healthy Male and Female Volunteers
Brief Title: Effects of Teduglutide on Cardiac Repolarisation and Conduction in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Head of Exploratory Clinical Development, Nycomed GmbH
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TE-1777-102-EC
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: Thorough QTc-Study; Short Bowel Syndrome; Cardiac safety
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Teduglutide 5 mg (Experimental): Treatment A, subcutaneous injection
  Interventions: Drug: Teduglutide
- Teduglutide 20 mg (Experimental): Treatment B, subcutaneous injection
  Interventions: Drug: Teduglutide
- Placebo (Placebo Comparator): subcutaneous injection
  Interventions: Drug: Teduglutide
- Moxifloxacin (Active Comparator): 400 mg, oral
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — subcutaneous (SC), single dose

SUMMARY:
The primary objective of this trial is to investigate if teduglutide has an effect on cardiac repolarisation (QT, QTc interval). Secondary objectives are the investigation of possible effects on heart rate and cardiac conduction (RR and PR intervals, QRS duration), pharmacokinetics and safety and tolerability in healthy subjects, and to determine the effect of the positive control, moxifloxacin, for sensitivity analysis. The trial will consist of a screening and a treatment phase of four treatment periods. There is a washout period of at least 7 days and 4 weeks at maximum between administrations. The expected total trial duration for the individual subject will be about 7 weeks (maximum 17) weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers
* Normal body weight (body mass index within ≥18 and 29 kg/m2 (inclusive) and a body weight >50 kg (females) and >60 kg (males).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
ECG measurement/assessment to determine the effect of a single dose of teduglutide on cardiac repolarisation (QT, QTc interval). | until 24 h post dose

SECONDARY OUTCOMES:
ECG measurement/assessment to determine the effect of a single dose of a positive control, moxifloxacin, on cardiac repolarisation, heart rate, and conduction | until 24 h post dose
ECG measurement/assessment to determine the effect of a single dose of teduglutide on heart rate and cardiac conduction (RR and PR intervals, QRS duration) | until 24 h post dose
PK blood samples to investigate pharmacokinetics of teduglutide in plasma | until 24 h post dose
PK blood samples to explore the concentration effect relationship on QT/QTc intervals | until 24 h post dose
ECG measurement/assessment and PK blood samples to investigate safety and tolerability of teduglutide | within 14 days after trial medication administration

CONTACTS AND LOCATIONS:
Locations (1):
- Nycomed GmbH, Konstanz, Germany